CLINICAL TRIAL: NCT01138410
Title: A Phase I/II Trial of SCIB1, a DNA Immunotherapy, in the Treatment of Patients With Malignant Melanoma
Brief Title: Study of a DNA Immunotherapy to Treat Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Product availability
Sponsor: Scancell Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCIB1-001
Record Dates: First submitted 2010-05-24; First posted 2010-06-07 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Malignant Melanoma
Keywords: Immunotherapy; Melanoma; Gene therapy; DNA plasmid; Cancer vaccine; Electroporation; CTL response
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCIB1 (Experimental)
  Interventions: Biological: SCIB1

INTERVENTIONS:
Biological: SCIB1 — Aqueous solution of plasmid DNA administered by intramuscular injection using the TDS-IM electroporation device (Ichor Medical Systems, Inc.) at week 0, 3, 6, 12 and 24. Part 1 of the study will escalate through 0.4, 2.0, 4.0 and 8.0 mg dose level cohorts, each of three patients. In Part 2 of the study the 4.0 and 8.0 mg doses will be administered in the same regimen. At the discretion of the investigator, patients in both parts of the study may continue to receive SCIB1 at 3-6 month intervals for 5 years.

SUMMARY:
The study is an investigation of a novel immunotherapy, SCIB1, for the treatment of melanoma. SCIB1 is a solution of plasmid DNA molecules which will express a modified antibody in human cells. The antibody modifications are designed to stimulate the patient's immune T cells to have a strong and specific reaction against melanoma cells which should then be eliminated. SCIB1 is injected into muscle using a device which simultaneously delivers an electrical impulse to enhance the transfer of SCIB1 into muscle cells. The trial will assess the safety and tolerability of SCIB1, the safety and performance of the injection device and the immunological effects of SCIB1. This is the first study of SCIB1 in humans and the trial has two parts, in the first part the dose will be escalated to determine a safe and tolerable level up to a maximum of 8 mg per dose. In the second part patients will receive the dose determined in the first part. Patients will have stage III or IV melanoma, be HLA type A2 and have a life expectancy of at least three months. All patients will receive 5 injections of SCIB1 over 5.5 months. At the discretion of the investigator, patients may continue to receive SCIB1 at 3-6 month intervals for 5 years. The study will be conducted at major cancer centres in the UK only and is expected to last for seven years. Patients will be followed up for five years after they have completed the trial.

ELIGIBILITY:
Inclusion Criteria:

Part One and Part Two (8.0 mg dose):

* Histologically confirmed Stage IV or Stage III malignant melanoma, as defined by the American Joint Committee on Cancer (AJCC).
* Must have measurable disease (RECIST 1.0)

Part Two (4.0 mg dose) only:

* Histologically confirmed, resected Stage III or resected Stage IV malignant melanoma, as defined by the AJCC, within 12 months of resection and with no tumour detectable at the time of screening.

Part One and Part Two:

* HLA-A2 positive.
* Positive for HLA-DR4, HLA-DR7, HLA-DR53 or HLA-DQ6.
* Lymphocyte count ≥ 5 x 10e9 cells/mL.
* Serum lactate dehydrogenase (LDH) ≤ upper limit of normal.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Willing and able to give written, informed consent.
* If male or female of childbearing potential, must be willing to use an effective contraceptive during the course of the study and for three months afterwards.

Exclusion Criteria:

* Known brain metastases at screening.
* Life expectancy of less than three months.
* Patients with TNM classification M1c at screening.
* Prior systemic anti-cancer treatment within four weeks of screening.
* Prior treatment with systemic corticosteroids or other immunosuppressants within four weeks of screening.
* Previous (within five years) or current malignancy at other sites with the exception of curatively treated local tumours such as carcinoma-in-situ of the cervix, basal or squamous cell carcinoma of the skin.
* Pregnant or lactating women.
* Presence of any uncontrolled and significant medical or psychiatric condition which would interfere with trial safety assessments. Caution should be used for patients with suspected or diagnosed epilepsy.
* Any electronic stimulation device such as cardiac demand pacemaker, automatic implantable cardiac defibrillator, nerve stimulators or deep brain stimulators.
* Individuals in which a skin-fold measurement of the cutaneous and subcutaneous tissue for all eligible injection sites (deltoid or quadriceps muscles with intact lymph drainage) exceeds 40 mm.
* Individuals with a heart rate of ≤ 50 beats per minute, history of significant cardiac abnormality and/or significant abnormal baseline electrocardiogram (ECG) readout.
* Treatment with any investigational product within the four weeks preceding screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability | Duration of treatment phase: up to 5.5 years
  Recording and assessment of adverse events to establish safety and tolerability of an investigational immunotherapy, SCIB1, in patients with melanoma whose cancer has spread from the initial tumour (i.e., stage III or stage IV melanoma).

SECONDARY OUTCOMES:
Safety, tolerability, biological and clinical effects | Duration of treatment phase: up to 5.5 years
  (i) Recording and assessment of adverse events and patient recorded experience to establish safety and tolerability of SCIB1 administered intramuscularly to melanoma patients using the TDS IM device.
  (ii) Cellular immune response by ex vivo assay induced by SCIB1 administered intramuscularly to melanoma patients using the TDS-IM device.
  (iii) Tumour response by CT scan in patients treated with SCIB1 (Part One only).

CONTACTS AND LOCATIONS:
Overall Officials: Poulam M Patel, MD, Study Director — Department of Clinical Oncology, City Hospital, Nottingham, UK; Paul Lorigan, MD, Principal Investigator — Department of Medical Oncology, Christie Hospital, Manchester, UK; Maria Marples, MD, Principal Investigator — St James' Institute of Oncology, Leeds, UK; Christian Ottensmeier, MD, Principal Investigator — Department of Medical Oncology, Southampton General Hospital, UK; Hardev Pandha, MD, Principal Investigator — Department of Medical Oncology, Royal Surrey County Hospital, Guildford, UK
Locations (5):
- United Kingdom (5):
  - Department of Medical Oncology, The Royal Surrey County Hospital, Guildford, Surrey
  - St James' Institute of Oncology, Leeds
  - Christie Hospital, Manchester
  - Department of Clinical Oncology, City Hospital, Nottingham
  - Department of Medical Oncology, Southampton General Hospital, Southampton